CLINICAL TRIAL: NCT03325608
Title: Program of Intensive Support in Emergency Departments for Care Partners of Cognitively Impaired Patients
Acronym: POISED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-01473; 1R01AG054574-01 (NIH)
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POISED Care (Experimental): Dyads randomized to the POISED Care intervention will work with the POISED care management team - consisting of specially-trained nurses functioning as care managers (CMs) and para-professionals in the role of care manager assistants (CMAs) - to create an individualized care plan through the lens of cognitive impairment with an emphasis on coordinating care with the patient's primary care provider (PCP) and achieving relevance with the goals and capacity of the family care-giver and care-recipient.
  Interventions: Other: POISED Care
- Usual Care (No Intervention): Participants will receive referrals to services at the time of enrollment.

INTERVENTIONS:
Other: POISED Care — Program of dementia care management.
  Arms: POISED Care

SUMMARY:
Dementia is a common problem for older patients presenting to emergency departments and for the family caregivers who often lack support, understanding, and skills to manage the problems related to the need for emergency department visits. The purpose of Program of Intensive Support in Emergency Departments for Care Partners of Cognitively Impaired Patients (POISED-CPCIP, here on referred to as POISED) randomized controlled trial is to use previously established quality improvement methods of root cause analysis to uncover reasons for emergency department use and to focus on caregiver activation within a program of dementia care management.

The goals of this study are to reduce recurrent emergency department visits and improve caregiver symptoms of depression, anxiety and need for social support.

ELIGIBILITY:
Inclusion Criteria:

* Must be in the emergency department for care at the point of recruitment
* Must be English- or Spanish-speaking
* Must have a family member or friend who provides caregiving assistance
* Must have a plan to be discharged to home (ESI = 4 or 5)
* Must have score <3 on the MiniCog or if using caregiver assessment by IQCODE must be >3.4
* Must have capacity to consent or have a proxy.

Exclusion Criteria:

* Care recipient (CR) is a resident of a nursing home or other supportive facility
* CR scores > 3 on the MiniCog or the caregiver assessment by IQCODE was < 3.4
* Caregiver (CG) declines participation
* CR is not being discharged to home

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 889 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Chodosh J, Connor K, Fowler N, Gao S, Perkins A, Grudzen C, Messina F, Mangold M, Smilowitz J, Boustani M, Borson S. Program of Intensive Support in Emergency Departments for Care Partners of Cognitively Impaired Patients: Protocol for a Multisite Randomized Controlled Trial. JMIR Res Protoc. 2022 Oct 20;11(10):e36607. doi: 10.2196/36607. PMID 36264626

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol enrollment of "889" represents the total number of patient/care-provider dyads; 247 dyads did not start the trial.
Groups:
- POISED Care Intervention - Patients: Participants assigned to the POISED Care Intervention. The POISED care management team consisting of specially-trained nurses functioning as care managers (CMs) and para-professionals in the role of care manager assistants (CMAs) will conduct a biopsychosocial/environmental needs assessment by phone within 48 hours of emergency room discharge if not possible during the ED stay.
  POISED Care: Using information collected, a propose plan of care and tailored interventions to the patients. Patients will understand natural history, and the prognosis of dementia; care protocols will be implemented.
- POISED Care Intervention - Caregivers of Patients: Caregivers of patients assigned to receive the POISED Care intervention.
- Usual Care - Patients: Patients will receive referrals to services at the time of enrollment.
  Usual Care: Usual care group will not receive the POISED structured assessment, attention to chronic disease management, or RCA related to the ED visit.
- Usual Care - Caregivers of Patients: Caregivers of patients assigned to receive usual care.
Period: Overall Study
Arm/Group | POISED Care Intervention - Patients | POISED Care Intervention - Caregivers of Patients | Usual Care - Patients | Usual Care - Caregivers of Patients
Started | 320 | 320 | 322 | 322
Completed | 207 | 207 | 222 | 222
Not Completed | 113 | 113 | 100 | 100
Not completed — Lost to Follow-up | 23 | 23 | 30 | 30
Not completed — Death of Caregiver | 0 | 0 | 2 | 2
Not completed — Death of Care Recipient | 34 | 34 | 28 | 28
Not completed — Withdrawal by Subject | 49 | 49 | 35 | 35
Not completed — Ineligible | 7 | 7 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- POISED Care Intervention - Care Givers of Patients: Caregivers of patients assigned to receive the POISED Care Intervention.
- Usual Care - Care Givers of Patients: Caregivers of patients assigned to receive usual care.
- Total: Total of all reporting groups
Arm/Group | POISED Care Intervention - Patients | POISED Care Intervention - Care Givers of Patients | Usual Care - Patients | Usual Care - Care Givers of Patients | Total
Number analyzed (Participants) | 320 | 320 | 322 | 322 | 1284
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.3 (6.3) | 60.9 (11.8) | 85.1 (6.1) | 59.6 (13.3) | 72.725 (9.375)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 221 | 230 | 201 | 240 | 892
  Male | 99 | 89 | 121 | 80 | 389
  Unknown or not reported | 0 | 1 | 0 | 1 | 2
  Prefer Not to Answer | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 58 | 33 | 69 | 188
  Not Hispanic or Latino | 188 | 261 | 184 | 251 | 884
  Unknown or Not Reported | 104 | 1 | 105 | 2 | 212
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 3 | 5
  Asian | 6 | 8 | 7 | 8 | 29
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 56 | 58 | 57 | 58 | 229
  White | 199 | 207 | 192 | 193 | 791
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 57 | 47 | 64 | 60 | 228
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 3 | 5
  Asian | 6 | 8 | 7 | 8 | 29
  Native Hawaiian or Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 56 | 58 | 57 | 58 | 229
  White | 199 | 207 | 192 | 193 | 791
  More than one race | 0 | 0 | 0 | 0 | 0
  Other | 0 | 43 | 0 | 56 | 99
  Unknown or not reported | 57 | 4 | 64 | 4 | 129
Region of Enrollment [Number; unit: participants]
  United States | 320 | 320 | 322 | 322 | 1284

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Emergency Department (ED) Visit Within 6 Months After Enrollment
Description: Percentage of participants who visit the ED within 6 months of being enrolled.
Time Frame: Up to Month 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | POISED Care Intervention - Patients | Usual Care - Patients
Number analyzed (Participants) | 315 | 317
percentage of participants | 41.60 [36.1 to 47.3] | 39.40 [34.0 to 45.1]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious and Other Adverse Events were not formally monitored/assessed among participants (patients and caregivers).
Groups:
- POISED Care Intervention - Care Givers of Patients: Caregivers of patients assigned to POISED Care intervention.
- Usual Care - Care Givers of Patients: Caregivers of patients assigned to usual care.
Arm/Group | POISED Care Intervention - Patients | POISED Care Intervention - Care Givers of Patients | Usual Care - Patients | Usual Care - Care Givers of Patients
All-Cause Mortality (participants affected / at risk) | 34/320 | 0/320 | 28/322 | 2/322
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03325608/Prot_SAP_000.pdf